CLINICAL TRIAL: NCT06793241
Title: A Clinical Study on the Safety and Effectiveness of Donor Derived CD19 CAR-T Cells in the Treatment of R/R B-cell Acute Lymphoblastic Leukemia
Brief Title: Donor Derived CD19 CAR-T Cells in the Treatment of R/R B-cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024011
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: CD19 CAR-T
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CD19 B-cell Acute Lymphoblastic Leukemia Targeted CAR T-cells (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CD19 B-cell Acute Lymphoblastic Leukemia Targeted CAR T-cells injection

INTERVENTIONS:
Biological: CD19 B-cell Acute Lymphoblastic Leukemia Targeted CAR T-cells injection — Each subject receive CD19 B-cell Acute Lymphoblastic Leukemia Targeted CAR T-cells by intravenous infusion

SUMMARY:
A Clinical Study on the Safety and Effectiveness of donor derived CD19 CAR-T Cells in the treatment of R/R B-cell acute lymphoblastic leukemia

DETAILED DESCRIPTION:
In this study, 15 patients with relapsed refractory B-cell acute lymphoblastic leukemia were proposed to undergo CD19 CAR-T Cells therapy. Under the premise that its safety has been clarified in previous studies, further observation and evaluation of the effectiveness of CD19 CAR-T Cells therapy for relapsed refractory B-cell acute lymphoblastic leukemia; At the same time, on the basis of expanding the sample size, more safety data on CD19 CAR-T Cells treatment for relapsed refractory B-cell acute lymphoblastic leukemia were accumulated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, gender unlimited;
* 2. Abnormal B cell immunotyping was CD19 positive;
* 3. Patients diagnosed with B-cell acute lymphoblastic leukemia by histological or immunotyping;
* 4. Meets the diagnosis of relapsed or refractory B-cell acute lymphoblastic leukemia (R/R B-ALL) and includes any of the following conditions:

  1. No CR was obtained after standard chemotherapy;
  2. CR was induced for the first time, but the duration of CR was less than 12 months;
  3. R/R B-ALL that does not work after the first or more remedial treatments;
  4. Two or more relapses;
* 5. The researchers believed that the patient had been adequately treated, such as auto-HSCT, auto-CART could not be prepared or preparation failed. Autologous CAR-T preparation failure was defined as including too few autologous lymphocytes (<1×109) or insufficient expansion during preparation or failure to meet the release criteria;
* 6. Total bilirubin ≤51 ( μmol/L), alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal, creatinine ≤176.8 (μmol/L);
* 7. Absolute neutrophil count: ≥ 0.5×109/L; Platelet: ≥ 30×109/L; Hemoglobin ≧60g/L;
* 8. Echocardiography showed left ventricular ejection fraction (LVEF) ≥40%;
* 9. The estimated survival is more than 3 months;
* 10. ECOG score 0-2;
* 11. Women and men who are fertile must consent to the use of appropriate contraception before entering the study, during study participation, and for 6 months after transfusion (the safety of this therapy for the unborn child is not known, with unknown risks);
* 12. Subjects who are willing to participate in the study are able to understand and have the ability to sign informed consent.

Exclusion Criteria:

* 1. Known allergies to research preconditioning measures, etc;
* 2. People with a history of epilepsy or other central nervous system disorders;
* 3. People with a history of prolonged QT or severe heart disease;
* 4. Less than 100 days after receiving allogeneic hematopoietic stem cell transplantation;
* 5. Hiv-infected person;
* 6. Persons with active hepatitis B or C virus; Those who are not cured have active infections;
* 7. Insufficient amplification ability (< 5x) in response to CD3 / CD28 costimulatory signals;
* 8. Combined use of systemic steroids (e.g., prednisone ≥20mg) within 3 days prior to screening, except for ongoing or intermittent use of topical, inhaled or intranasal steroids within 2 weeks or at present; Or have systemic diseases that require long-term use of immunological agents;
* 9. Patients who received anti-cancer chemotherapy or other drugs within 2 weeks prior to screening;
* 10. Any situation that the investigator believes may increase the risk of the subjects or interfere with the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Duration of remission ,DOR | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Overall survival, OS | Up to 2 years after Treatment
  After transplantation until death from any cause.
Event-free survival (EFS) | Up to 1 years after CAR-T infusion
  defined as the time from the date of receiving the infusion to the date of treatment failure (failure to achieve CR/CRh/CRi/MLFS/PR after both efficacy assessments), or relapse (hematologic relapse or extramedullary relapse after CR/CRh/CRi), or death from any cause, whichever occurs first. When an EFS event was "Ineffective Therapy", the primary analysis of EFS was performed on a 1-day basis (ie, time to treatment received as the event). For a more comprehensive assessment, sensitivity analyses could be performed using the actual date of treatment failure, end of treatment, or start of next-line anti-leukemia therapy as the end of EFS for treatment failure, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China